CLINICAL TRIAL: NCT00835068
Title: Post Marketing Observational Study Of Reformulated BeneFIX
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 3090X1-4409; B1821007
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Results first posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Hemophilia B
Keywords: Hemophilia B; observational; post marketing study
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BeneFIX
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — As it is a non interventional study, patient receives his usual treatment (BeneFIX) as determined by the physician

SUMMARY:
The primary objective of this observational study is to collect safety data on reformulated BeneFIX as prescribed in routine clinical practice conditions in France. The secondary objectives are to collect data on the clinical course of individuals treated with reformulated BeneFIX and on the ease of reformulated BeneFIX.

DETAILED DESCRIPTION:
No sampling

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Hemophilia B already receiving or starting treatment with reformulated BeneFIX.
* Subjects who have dated and signed the informed consent form.

Exclusion Criteria:

* Ongoing treatment of Hemophilia B by a product other than reformulated BeneFIX.
* Participation in the European prospective registry of patients with Hemophilia B treated with BeneFIX (Wyeth protocol 3090A-101039).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hemophilia B patients already receiving or starting treatment with reformulated BeneFIX
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2009-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- France (16):
  - Pfizer Investigational Site, Chamberry, Cedex
  - Pfizer Investigational Site, Le Chesnay, Cedex
  - Pfizer Investigational Site, Caen
  - Pfizer Investigational Site, Clermont-Ferrand
  - Pfizer Investigational Site, Dijon
  - Pfizer Investigational Site, leKremlin-Bicetre
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Montmorency
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Nantes
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Rouen
  - Pfizer Investigational Site, Saint-Priest-en-Jarez
  - Pfizer Investigational Site, Tours
  - Pfizer Investigational Site, Vandœuvre-lès-Nancy

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3090X1-4409&StudyName=Post%20Marketing%20Observational%20Study%20of%20reformulated%20BeneFIX

RESULTS

PARTICIPANT FLOW:
Groups:
- BeneFIX (Previously Treated Participants): Participants with hemophilia B who were previously treated with reformulated BeneFIX, received reformulated BeneFIX intravenous injection per routine clinical practice and were observed for up to 5 years.
- BeneFIX (Previously Untreated Participants): Participants with hemophilia B who were previously untreated with reformulated BeneFIX, received reformulated BeneFIX intravenous injection as per routine clinical practice and were observed for up to 5 years.
Period: Overall Study
Arm/Group | BeneFIX (Previously Treated Participants) | BeneFIX (Previously Untreated Participants)
Started | 57 | 1
Completed | 47 | 0
Not Completed | 10 | 1
Not completed — Death | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Other | 8 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of BeneFIX.
Groups:
- Total: Total of all reporting groups
Arm/Group | BeneFIX (Previously Treated Participants) | BeneFIX (Previously Untreated Participants) | Total
Number analyzed (Participants) | 57 | 1 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.36 (16.237) | 1.30 | 22.98 (16.353)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 57 | 1 | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Related Adverse Events (AEs) and Serious Adverse Events (SAEs) Prior to Safety Amendment
Description: A treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included SAEs as well as non-serious AEs which occurred prior to safety amendment. Prior to safety amendment, only AEs/SAEs deemed related to BeneFIX as per participating physician were collected.
Time Frame: Baseline up to Year 3.5
Population: Safety population included all participants who received at least one dose of BeneFIX.
Measure: Number; unit: participants
Arm/Group | BeneFIX (Previously Treated Participants) | BeneFIX (Previously Untreated Participants)
Number analyzed (Participants) | 57 | 1
participants
  Treatment-related AE | 1 | 1
  Treatment-related SAE | 0 | 1

2. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) by Relationship After Safety Amendment
Description: AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. A treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug as per participating physician. AEs included SAEs as well as non-serious AEs which occurred after the safety amendment. After the safety amendment, all AEs/SAEs were collected irrespective of their relationship to BeneFIX.
Time Frame: Year 3.5 up to 4.75
Population: Safety population included all participants who received at least one dose of BeneFIX. Previously untreated participants were not evaluable for this outcome measure due to discontinuation prior to safety amendment.
Measure: Number; unit: participants
Arm/Group | BeneFIX (Previously Treated Participants) | BeneFIX (Previously Untreated Participants)
Number analyzed (Participants) | 57 | 0
participants
  AE | 26 |
  SAE | 10 |
  Treatment-related AE | 1 |
  Treatment-related SAE | 0 |

3. Primary Outcome: Number of Participants With Events of Special Interest
Description: Events of special interest included allergic reactions, red blood cell (RBC) agglutination phenomena, lack of efficacy/low recovery, thrombotic events and onset of factor IX (FIX) inhibitor. Participants may be represented in more than 1 category.
Time Frame: Baseline up to Year 4.75
Population: Safety population included all participants who received at least one dose of BeneFIX.
Measure: Number; unit: participants
Arm/Group | BeneFIX (Previously Treated Participants) | BeneFIX (Previously Untreated Participants)
Number analyzed (Participants) | 57 | 1
participants
  FIX inhibitor | 0 | 1
  Allergic reactions | 0 | 0
  RBC agglutination | 0 | 0
  Lack of efficacy/ low recovery | 0 | 0
  Thrombotic event | 0 | 0

4. Secondary Outcome: Number of Bleeding Episodes
Description: Number of bleeding episode during prophylaxis and on demand period were reported. All periods with at least one injection per week were considered as prophylaxis period. All prophylaxis periods of less than a month were reviewed and cross-checked with the treatment scheme planned at the previous visit to confirm if they were real prophylaxis periods or preventive injections periods. On demand treatment period included the total duration of follow up excluding duration of both prophylaxis and preventive injection treatment scheme. Efficacy population included only those participants who were previously treated with BeneFIX. Here, 'n' signifies participants evaluable for this measure during the specified treatment period. Participants may be represented in more than 1 category.
Time Frame: Baseline up to Year 4.75
Population: Efficacy population: participants with basal FIX activity less than or equal to (<=) 1 percent (%) with real exposure days in diary at least 70% of planned exposure days for prophylaxis period, and without FIX inhibitor before or during study (no FIX inhibitor history at baseline; FIX inhibitor titer <0.6 Bethesda Unit [BU] during follow up).
Measure: Number; unit: bleeding episodes
Arm/Group | BeneFIX (Previously Treated Participants)
Number analyzed (Participants) | 42
bleeding episodes
  Prophylaxis (n=28) | 261
  On demand (n=21) | 695

5. Secondary Outcome: Number of Bleeding Episodes Requiring Treatment by Injection
Description: Number of injections (1, 2, 3 or greater than or equal to [>= 4]) required to treat the bleeding episodes during prophylaxis and on demand period were reported. All periods with at least one injection per week were considered as prophylaxis period. All prophylaxis periods of less than a month were reviewed and cross-checked with the treatment scheme planned at the previous visit to confirm if they were real prophylaxis periods or preventive injections periods. On demand treatment period included the total duration of follow up excluding duration of both prophylaxis and preventive injection treatment scheme.
Time Frame: Baseline up to Year 4.75
Population: Efficacy population. Efficacy population included only those participants who were previously treated with BeneFIX. Here, 'number of bleeding episodes analyzed' signifies episodes evaluable for this measure. 'n' signifies those bleeding episodes with injection data available during specified period.
Measure: Number; unit: bleeding episodes
Units Other Than Participants: bleeding episodes
Arm/Group | BeneFIX (Previously Treated Participants)
Number analyzed (Participants) | 42
Number analyzed (bleeding episodes) | 955
bleeding episodes
  Prophylaxis: 1 Injection (n = 261) | 144
  On demand: 1 Injection (n = 694) | 515
  Prophylaxis: 2 Injection (n = 261) | 63
  On demand: 2 Injection (n = 694) | 89
  Prophylaxis: 3 Injection (n = 261) | 21
  On demand: 3 Injection (n = 694) | 35
  Prophylaxis: >=4 Injection (n = 261) | 33
  On demand: >=4 Injection (n = 694) | 55

6. Secondary Outcome: Total Consumption of BeneFIX
Description: Total consumption of BeneFIX included consumption during prophylaxis, on demand, during bleeding episodes, preventive injections, surgeries or immune tolerance.
Time Frame: Baseline up to Year 4.75
Population: Safety population included all participants who received at least one dose of BeneFIX. Participants with at least one follow-up visit were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: International Unit (IU)
Arm/Group | BeneFIX (Previously Treated Participants) | BeneFIX (Previously Untreated Participants)
Number analyzed (Participants) | 51 | 1
International Unit (IU) | 434751.0 (446077.9) | 15000.0

7. Secondary Outcome: Subjective Assessment of Efficacy by Participant
Description: Participants assessed efficacy of BeneFIX as very good, good, moderate and bad at each follow-up visit. Results were summarized for the latest (most recent), worst and best assessment of BeneFIX done by the participant.
Time Frame: Baseline up to Year 4.75
Population: Efficacy population. Efficacy population included only those participants who were previously treated with BeneFIX.
Measure: Number; unit: participants
Arm/Group | BeneFIX (Previously Treated Participants)
Number analyzed (Participants) | 42
participants
  Latest assessment: Missing Values | 4
  Latest assessment: Very Good | 19
  Latest assessment: Good | 19
  Latest assessment: Moderate | 0
  Latest assessment: Bad | 0
  Worst assessment: Missing Values | 4
  Worst assessment: Very Good | 17
  Worst assessment: Good | 20
  Worst assessment: Moderate | 1
  Worst assessment: Bad | 0
  Best assessment: Missing Values | 4
  Best assessment: Very Good | 25
  Best assessment: Good | 13
  Best assessment: Moderate | 0
  Best assessment: Bad | 0

8. Secondary Outcome: Dose Per Injection of BeneFIX
Description: Dose per injection during prophylaxis and on demand period were reported. All periods with at least one injection per week were considered as prophylaxis period. All prophylaxis periods of less than a month were reviewed and cross-checked with the treatment scheme planned at the previous visit to confirm if they were real prophylaxis periods or preventive injections periods. On demand treatment period included the total duration of follow up excluding duration of both prophylaxis and preventive injection treatment scheme. Participants may be represented in more than 1 category.
Time Frame: Baseline up to Year 4.75
Population: Efficacy population. Efficacy population included only those participants who were previously treated with BeneFIX. Here, 'n' signifies participants evaluable for this measure during the specified treatment period.
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | BeneFIX (Previously Treated Participants)
Number analyzed (Participants) | 42
IU/kg
  Prophylaxis (n=28) | 45.3 (11.41)
  On demand (n=21) | 49.0 (14.25)

9. Secondary Outcome: Subjective Assessment of Efficacy by Physician
Description: Participating physician assessed efficacy of BeneFIX as very good, good, moderate and bad at follow-up visit. Results were summarized for the latest (most recent), worst and best assessment of BeneFIX done by the physician.
Time Frame: Baseline up to Year 4.75
Population: Efficacy population. Efficacy population included only those participants who were previously treated with BeneFIX.
Measure: Number; unit: participants
Arm/Group | BeneFIX (Previously Treated Participants)
Number analyzed (Participants) | 42
participants
  Latest assessment: Very Good | 17
  Latest assessment: Good | 23
  Latest assessment: Moderate | 2
  Latest assessment: Bad | 0
  Worst assessment: Very Good | 10
  Worst assessment: Good | 29
  Worst assessment: Moderate | 3
  Worst assessment: Bad | 0
  Best assessment: Very Good | 31
  Best assessment: Good | 11
  Best assessment: Moderate | 0
  Best assessment: Bad | 0

10. Secondary Outcome: Subjective Assessment of Ease of Use by Participant
Description: Participants assessed ease of use of BeneFIX as very good, good, moderate and bad at each follow-up visit. Results were summarized for the latest (most recent), worst and best assessment of BeneFIX done by the participant.
Time Frame: Baseline up to Year 4.75
Population: Efficacy population. Efficacy population included only those participants who were previously treated with BeneFIX.
Measure: Number; unit: participants
Arm/Group | BeneFIX (Previously Treated Participants)
Number analyzed (Participants) | 42
participants
  Latest assessment: Missing | 5
  Latest assessment: Very Good | 17
  Latest assessment: Good | 19
  Latest assessment: Moderate | 1
  Latest assessment: Bad | 0
  Worst assessment: Missing Value | 5
  Worst assessment: Very Good | 13
  Worst assessment: Good | 22
  Worst assessment: Moderate | 2
  Worst assessment: Bad | 0
  Best assessment: Missing Values | 5
  Best assessment: Very Good | 21
  Best assessment: Good | 16
  Best assessment: Moderate | 0
  Best assessment: Bad | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | BeneFIX (Previously Treated Participants) | BeneFIX (Previously Untreated Participants)
Serious Adverse Events (participants affected / at risk) | 10/57 | 1/1
Other Adverse Events (participants affected / at risk) | 21/57 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BeneFIX (Previously Treated Participants) (N=57) | BeneFIX (Previously Untreated Participants) (N=1)
Factor IX inhibition (Blood and lymphatic system disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Device failure (General disorders) | 1 | 0
Hyperthermia (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Otitis media (Ear and labyrinth disorders) | 1 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0
Congenital genitourinary abnormality (Congenital, familial and genetic disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BeneFIX (Previously Treated Participants) (N=57) | BeneFIX (Previously Untreated Participants) (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Branchial cyst (Congenital, familial and genetic disorders) | 1 | 0
Ear infection (Ear and labyrinth disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Mucosal dryness (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Varicella (Infections and infestations) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Vitamin D increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Speech disorder (Nervous system disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Haematospermia (Reproductive system and breast disorders) | 1 | 0
Asthma exercise induced (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Vascular disorders) | 1 | 0
Haemorrhoids (Vascular disorders) | 2 | 0
Rectal haemorrhage (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.